CLINICAL TRIAL: NCT03499288
Title: A Multi-country, Multi-centre, Observational, Cross-sectional Study to Evaluate Individualized Treatment and Management in Children and Adolescents With Cerebral Palsy
Brief Title: Profiling Children and Youth With Cerebral Palsy in Relation to Feeding and Nutrition
Acronym: Purple-N
Status: Completed | Type: Observational
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Other Study IDs: MPR15FA89628
Record Dates: First submitted 2018-03-21; First posted 2018-04-17 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and youth with cerebral palsy: Subjects between 1 month and 18 years of age with Cerebral Palsy who visited the coordinating HCP within the past 12 months.

SUMMARY:
HCPs will complete questionnaires about their patients with Cerebral Palsy (CP) and invite parents/caregivers of these patients to fill in questionnaires as well. Questionnaires include questions on individualized treatment, nutritional profile and management, and patient characteristics.

DETAILED DESCRIPTION:
Coordinating health care professionals (HCPs; e.g. paediatric neurologists, physiotherapists) in different centres across different countries will be asked to participate in this cross-sectional study.

A) for the HCP to fill out a questionnaire about their CP child, related to general subject characteristics, motor function, co-morbidities, type of therapies, anthropometry, feeding mode and nutritional status; and B) for parents (/legal representatives) to receive and fill out questionnaires about their CP child and themselves, related to general subject characteristics, motor function, co-morbidities, type of therapies, anthropometry, feeding mode and nutritional status, participation and (their own) quality of life.

If parents (/legal representatives) agree to "A)", but not "B)" then a subject will still enter the study, but without the parental assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Cerebral Palsy
2. Age<18 years
3. Have visited the HCP within the last year
4. Written informed consent provided by parents/legal representatives according to local law

Exclusion Criteria:

1. Neurodegenerative diseases
2. Acute infections: meningitis, encephalitis or poliomyelitis

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects between 1 month and 18 years of age with Cerebral Palsy
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Quantify current CP characteristics 1 (general subject characteristics): | Data collected retrospectively, from within 12 months of entering the questionnaire
  Using questionnaires to quantify current CP characteristics with respect to:
  - General subject characteristics (e.g. Sex, Birth weight [g], Type of CP motor disorder [category]
Quantify current CP characteristics 2 (anthropometry): | Data collected retrospectively, from within 12 months of entering the questionnaire
  Using questionnaires to quantify current CP characteristics with respect to:
  Anthropometry: length [cm]; weight [grams] and BMI (kg/m2)
Quantify current CP characteristics 3 (motor function) | Data collected retrospectively, from within 12 months of entering the questionnaire
  Using questionnaires to quantify current CP characteristics with respect to:
  Motor function (GMFCS [category]; GMFM measurement type [GMFM-86/GMFM-88]
Quantify current CP characteristics 4 (comorbidities) | Data collected retrospectively, from within 12 months of entering the questionnaire
  Using questionnaires to quantify current CP characteristics with respect to:
  Comorbidities: epilepsy, cognitive function, GI problems [categories]
Quantify current CP characteristics 5 (therapies) | Data collected retrospectively, from within 12 months of entering the questionnaire
  Using questionnaires to quantify current CP characteristics with respect to:
  Type and frequency of physical/occupational therapy [type, number of hours per day /days per week]
Quantify current CP characteristics 6 (feeding mode) | Data collected retrospectively, from within 12 months of entering the questionnaire
  Using questionnaires to quantify current CP characteristics with respect to:
  Feeding mode and/or problems (tube feeding [yes/no], type of tube feeding etc)
Quantify current CP characteristics 7 (nutritional status) | Data collected retrospectively, from within 12 months of entering the questionnaire
  Using questionnaires to quantify current CP characteristics with respect to:
  Nutritional status (HCP and parent perspective on nutritional status, concerns [yes/no])

OTHER OUTCOMES:
Quality of life and participation 1 | Data collected retrospectively, from within 12 months of entering the questionnaire
  Questionnaire to assess Quality of Life of subjects with CP [scores on domains]
Quality of life and participation 2 | Data collected retrospectively, from within 12 months of entering the questionnaire
  Questionnaire to assess Quality of Life of parents (/legal representatives) of subjects with CP [scores on domains]
Quality of life and participation 3 | Data collected retrospectively, from within 12 months of entering the questionnaire
  Level of participation included in the general parent questionnaire [categories]

CONTACTS AND LOCATIONS:
Locations (20):
- Fakultní nemocnice v Motole, Prague, Czechia
- Attikon University General Hospital, Athens, Greece
- Bethesda Children Hospital Budapest, Budapest, Hungary
- Italy (4):
  - AO Sant'Orsola - Malpighi, Policlinico, Bologna
  - ASST degli Spedali Civili di Brescia, Brescia
  - Fondazione IRCCS Istituto Neurologico "Carlo Besta", Milan
  - AOU di Modena - Policlinico, Modena
- Roessingh centrum voor Revalidatie, Enschede, Netherlands
- Poland (2):
  - Medical university hospital of Gdansk, Gdansk
  - Szpital Kliniczny im. Heliodora Święcickiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
- Fakultná nemocnica Trnava, Trnava, Slovakia
- Turkey (Türkiye) (9):
  - Ankara University School of Medicine/Neurology, Ankara
  - Gazi University School of Medicine/Neurology, Ankara
  - Hacettepe University School of Medicine/Neurology, Ankara
  - Ege University School of Medicine/Neurology, Ege
  - Eskisehir Osmangazi University School of Medicine/Neurology, Eskişehir
  - Dokuz Eylul University School of Medicine/Neurology, Izmir
  - Inonu University School of Medicine/Neurology, İnönü
  - Marmara University School of Medicine/Neurology, Marmara
  - Mersin University School of Medicine/Neurology, Mersin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fogarasi A, Fazzi E, Smorenburg ARP, Mazurkiewicz-Beldzinska M, Dinopoulos A, Pobiecka A, Schroder-van den Nieuwendijk D, Kraus J, Tekgul H; PURPLE N study group; Czech Republic:; Kraus J; Greece:; Dinopoulos A, Koutsaki M; Hungary:; Fogarasi A; Italy:; Baranello G, Bertoli S, Caramaschi E, Cordelli DM, De Amicis R, Fazzi E, Forchielli ML, Guerra A, Lividini A, Marchio M, Rossi A; Netherlands:; Nieuwendijk DSD; Poland:; Flicinski J, Gurda B, Lemska A, Matheisel A, Mazurkiewicz-Beldzinska M, Niwinska Z, Pawlowicz M, Sawicka A, Steinborn B, Szmuda M, Winczewska-Wiktor A, Zawadzka M; Slovakia:; Pobiecka A; Turkey:; Arhan E, Aydin K, Bayram E, Carman KB, Edem P, Ertem D, Goktas OA, Gungor S, Haliloglu G, Kansu A, Komur M, Mutlu A, Kirsaclioglu CT, Okuyaz C, Ozgor B, Ozturk Y, Sager SG, Sarigecili E, Selimoglu MA, Serin HMO, Teber ST, Tekgul H, Thomas G, Turkdogan D, Volkan B, Yarar C, Yilmaz SK. The PURPLE N study: objective and perceived nutritional status in children and adolescents with cerebral palsy. Disabil Rehabil. 2022 Nov;44(22):6668-6675. doi: 10.1080/09638288.2021.1970255. Epub 2021 Sep 2. PMID 34473588